CLINICAL TRIAL: NCT01121965
Title: Early Vitrectomy for Impending Macular Hole. Multicenter Clinical Trial
Brief Title: Early Vitrectomy for Impending Macular Hole
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul Retina Investigator Group (Network)
Responsible Party: Se Woong Kang, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRIG #1
Record Dates: First submitted 2010-04-30; First posted 2010-05-12 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Retinal Perforation
Keywords: macular hole; impending macular hole; stage 1 macular hole
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conservative treatment group (No Intervention): Eyes which do not undergo early vitrectomy at the time of enrollment. Surgical intervention would be performed when full-thickness macular hole occurs
- Early vitrectomy (Experimental): Pars plana vitrectomy with ILM peeling would be employed when visual symptoms occur.
  Interventions: Procedure: Pars plana vitrectomy with ILM peeling

INTERVENTIONS:
Procedure: Pars plana vitrectomy with ILM peeling — Pars plana vitrectomy with ILM peeling
  Other Names: macular hole surgery
  Arms: Early vitrectomy

SUMMARY:
This study is designed to verify hypothesis that early vitrectomy may prevent impending macular hole from progression to full-thickness macular hole.

DETAILED DESCRIPTION:
In a study conducted 15 years ago, the 'Vitrectomy for Prevention of Macular hole Study Group' was not able to prove the benefits and advantages of vitrectomy for impending macular hole; however, during the interim period, notable improvements have been achieved with regard to diagnosis and efficacy of treatment.

Therefore, we designed this study to identify the effect of current vitreous surgery for symptomatic impending macular hole.

Characteristics of this study is as below

* Multicenter, prospective clinical trial. (early surgical intervention vs.surgical intervention when full-thickness macular hole occurs)
* Non-randomized study (decision was made by patients after full explanation)
* After 1 year follow up, functional change(visual acuity)and anatomical change(development of full-thickness macular hole) would be evaluated

ELIGIBILITY:
Inclusion Criteria:

* male or female with impending macular hole(identified with OCT)
* Age: over 45 years
* Symptom duration < 6 Months
* Visual acuity on trial: less than 73 letters in ETDRS chart Visual acuity of worsened eye: over 24 letters in ETDRS chart

Exclusion Criteria:

* Any vision disturbing disease other than impending macular hole
* Diabetic maculopathy or other retinal vascular disease
* Prior history of major trauma: If symptom begins after trauma
* Myopia over -6.5Dioper or eyes with axial length > 28mm
* Evidence of scar, degeneration or exudation of macula
* active intraocular inflammation
* History of intraocular surgery other than uncomplicated cataract extraction 3months before
* Uncontrolled IOP > 25mmHg

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual acuity | 48 weeks

SECONDARY OUTCOMES:
Rate of occurrence of full-thickness macular hole | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Se Woong Kang, M.D., Principal Investigator — Seoul Retina Investigator Group
Locations (10):
- South Korea (10):
  - Asan Medical Center, University of Ulsan College of Medicine, Seoul, 82-2-3010-3673
  - Konyang University, Myung Gok Eye Research Institute, Daejeon, Daejeon
  - Seoul National University Bundang Hospital, Seongnam, Gyunggi-do
  - HanGil Eye Hospital, Incheon, In Cheon
  - Seoul National University Hospital, Seoul, Seoul
  - Kangdong Sacred Heart Hospital, Hallym University College of Medicine,, Seoul, Seoul
  - Samsung Medical Center, Seoul, Seoul
  - Catholic University of Korea, Seoul, Seoul
  - Gangnam Sacred Heart Hospital,Hallym University, Seoul, Seoul
  - Kong eye clinic, Seoul, Seoul